CLINICAL TRIAL: NCT03160976
Title: Effects of Cryolipolysis on Localized Adiposity: Randomized Clinical Trial
Brief Title: Cryolipolysis on Localized Adiposity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECLA2017
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Subcutaneous Fat

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Subjects will only receive the Evaluation Protocol and will be followed for 90 days.
- Intervention Group (Active Comparator): A single 50 minutes session of cold exposure with a cryolipolysis device. The parameters will be: temperature -10°C and vacuum between 60 Kpas (at beginning) and 40 Kpas (until the end).
  Interventions: Other: Cryolipolysis

INTERVENTIONS:
Other: Cryolipolysis — First, the demarcation of the lower abdomen area at the same landmarks of the ultrasonography will be done. Secondly, the patient will be positioned on the stretcher in the supine position with a 45 ° elevation of the trunk. In this position, to protect the region to be treated, a glycerine antifreeze membrane will be placed. The treatment parameters will be: temperature of -10 ° C, treatment time of 50 minutes (first 3 minutes of heating at 42°C) and moderate vacuum pressure (60 - 40 Kpas). The applicator will be chosen according to the size of the area of each subject and positioned in the target region. At the end the skinfold will be released automatically, the antifreeze membrane removed and a manual massage will be carried out for five minutes to stimulate local blood reperfusion.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to analyze the effects of a single session of cryolipolysis on localized adiposity on women's abdomen. This is a randomized controlled clinical trial that will include 28 women who will be randomly allocated into two groups: Control Group or Intervention Group. The following assessments will be performed in both groups: ultrasonography and body composition at baseline and 30, 60 and 90 days after randomization and blood analysis at baseline and 15 and 30 days after randomization. The expected main result at the end of this study is the reduction of the local subcutaneous fat tissue.

DETAILED DESCRIPTION:
Cryolipolysis is a non - invasive method for localized fat reduction wich uses low temperatures to induce an apoptotic and inflammatory response and consequent adipocyte death in the treated area. Although the practice of this technique has been increasing, there are some gaps in the literature about the exact mechanism of action and only a few randomized clinical trials that proves its effectiveness and safety. Then, the aim of this study is to analyse the effects of cryolipolysis on localized fat on women's abdomen. This is a randomized controlled clinical trial that will include 28 women who will be randomized to Control Group (CG) or Intervention Group (IG). The CG will perform the Evaluation Protocol with the following assessments: ultrasonography, thermographic analysis, blood analysis, bioimpedance and measurement of skinfold and abdominal circumference. The IG will receive a single cryolipolysis's session on lower abdomen and the Evaluation Protocol. The follow up for both groups is 90 days. Expected main result at the end of the study is the reduction of the local subcutaneous fat tissue.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 to 45 or not being on menopause
* Sedentary according to International Physical Activity Questionnaire
* Body Mass Index lower than 27 Kg/m²
* Skinfold: more than 3 centimeters at the lower abdomen

Exclusion Criteria:

* Cryoglobulinemia
* Cold urticaria
* Paroxysmal cold hemoglobinuria
* Raynaud disease
* Pregnancy and Breastfeeding
* Cancer
* Vascular diseases
* Heart diseases
* Epidermal lesions at the site of application
* Autoimmune diseases
* Osteoporosis
* Metallic implants and pacemaker
* Alterations of sensibility
* Inflammatory process and active infection
* Abdominal hernia
* Abdominal muscle diastasis
* Diabetes
* Anemia
* Previous plastic surgery on the area
* Liver and kidney diseases
* Cognitive impairment that prevents conducting evaluations, as well as inability to understand and sign the informed consent form

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2017-05-25 (Estimated); Primary Completion 2017-08-25 (Estimated); Study Completion 2017-10-25 (Estimated)

PRIMARY OUTCOMES:
Subcutaneous fat layer | Baseline, 30, 60 and 90 days after intervention.
  Subcutaneous fat layer changes measured by ultrasonography and skinfold.

SECONDARY OUTCOMES:
Abdominal circumference | Baseline, 30, 60 and 90 days after intervention.
  Abdominal circumference changes measured by perimetry method.
Inflammatory profile | Baseline, 15 and 30 days after intervention.
  Inflammatory profile analyzed through level of interleukin - 6, tumor necrosis factor - alfa, monocyte chemotactic protein-1 and leptin.
Body fat mass | Baseline, 30, 60 and 90 days after intervention.
  Body fat mass changes measured by bioimpedance.
Liver function | Baseline, 15 and 30 days after intervention.
  Liver function analyzed through aspartate aminotransferase and alanine aminotransferase
Kidney function | Baseline, 15 and 30 days after intervention.
  Kidney function analyzed through creatinine and urea
Lipids profile | Baseline, 15 and 30 days after intervention
  Lipids profile analyzed through high density lipoprotein, low density lipoprotein, cholesterol, triglycerides and glucose levels.
Local temperature | 2 minutes before and 2 minutes after intervention and massage
  Local temperature changes with cryolipolysis measured by thermographic analysis.
Adverse effects | 15 days after intervention
  Identification of possible adverse effects by patient report
Pain level | First minute, twenty-fifth minute, fiftieth minute after intervention and first minute during the massage
  Pain level measured by analogue visual pain scale
Body weight and body mass index | Baseline, 30, 60 and 90 days after intervention.
  Body weight and body mass index
Physical Activity | Baseline and every 15 days after intervention
  Level of physical activity measured by the International Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Federal University of Health Science of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falster M, Schardong J, Santos DPD, Machado BC, Peres A, Rosa PVD, Plentz RDM. Effects of cryolipolysis on lower abdomen fat thickness of healthy women and patient satisfaction: a randomized controlled trial. Braz J Phys Ther. 2020 Sep-Oct;24(5):441-448. doi: 10.1016/j.bjpt.2019.07.005. Epub 2019 Jul 26. PMID 31375459